CLINICAL TRIAL: NCT04343157
Title: UCSD Image-Guided Cognitive-Sparing Radiosurgery for Brain Metastases: Avoidance of Eloquent White Matter and Hippocampal Regions
Brief Title: UCSD Image-Guided Cognitive-Sparing Radiosurgery for Brain Metastases
Acronym: IG-SRS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jona Hattangadi-Gluth (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jona Hattangadi-Gluth, Associate Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170848; R01CA238783-01 (NIH)
Record Dates: First submitted 2019-08-02; First posted 2020-04-13 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Brain Metastases, Adult; Neurocognitive Function; Cancer
MeSH Terms: conditions — Brain Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Study patients will undergo MR imaging with DTI and 3D volumetric imaging at baseline (pre-SRS), and 1 month, 3 months, and 6 months afterwards. This regimen of post-SRS MR imaging is clinical standard of care. Segmentation of critical white matter and hippocampal volumes will be performed pre-SRS for use in brain SRS planning. Formal neurocognitive assessments will be performed at baseline and 3 months post-SRS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Image-guided cognitive sparing brain SRS (Experimental): This is a single arm phase II study where enrolled subjects will receive intracranial SRS will performed identically to standard of care, except for implementing additional imaging techniques and software for additional regional avoidance for cognitive sparing (specifically sparing white matter and the bilateral hippocampus)
  Interventions: Radiation: Cognitive Sparing Brain Stereotactic Radiosurgery (SRS)

INTERVENTIONS:
Radiation: Cognitive Sparing Brain Stereotactic Radiosurgery (SRS) — In this proposal, the investigators introduce advanced diffusion and volumetric imaging techniques along with innovative, automated image parcellation methods to identify critical brain regions, incorporate into cognitive-sparing SRS, and analyze biomarkers of radiation response. This work will advance the investigators' understanding of neurocognitive changes after brain SRS and help create interventions that preserve cognitive-function in brain metastases patients.

SUMMARY:
In this proposal, the investigators introduce advanced diffusion and volumetric imaging techniques along with innovative, automated image parcellation methods to identify critical brain regions, incorporate into cognitive-sparing SRS, and analyze biomarkers of radiation response. This work will advance the investigators' understanding of neurocognitive changes after brain SRS and help create interventions that preserve cognitive-function in brain metastases patients.

DETAILED DESCRIPTION:
Background: Brain metastases affect one third of adult cancer patients. Stereotactic radiosurgery (SRS) is standard of care for patients with limited brain metastases. Yet most patients will experience post-treatment cognitive decline given the potential for high doses to eloquent white matter and the hippocampus.

Objective/Hypothesis: The investigator's team has developed innovative, robust imaging methods and automated segmentation techniques to identify critical white-matter tracts and the hippocampus using advanced diffusion tensor imaging (DTI) and volumetric imaging. These novel imaging techniques also allow us to directly and non-invasively measure microstructural changes after RT to critical brain structures in vivo. The investigators will use these advanced imaging technologies in a prospective trial of cognitive-sparing brain SRS for brain metastases patients.

Specific Aims: 1: To evaluate whether relative sparing of eloquent white matter tracts (critical for memory, language, attention, and executive functioning) and hippocampi from high doses during brain SRS results in improved 3-month post-SRS cognitive performance relative to historical controls in patients with 1 to 3 brain metastases. 2: To measure longitudinal trends in white matter damage (using DTI) and hippocampal atrophy (using volumetric change) among patients receiving cognitive-sparing brain SRS and correlate these imaging biomarkers with domain-specific cognitive outcomes.

Study Design: The investigators will prospectively enroll 60 adult patients with 1-3 brain metastases who are eligible for brain SRS and MRI. Patients will undergo MRI with DTI and 3D volumetric imaging at baseline (pre-SRS) and 1 month, 3 months, and 6 months afterwards. White matter and hippocampal segmentation will be performed and critical regions integrated into cognitive-sparing brain SRS planning with automated knowledge-based optimization. Cognitive-sparing dose constraints are derived from previous data. A well-established, validated battery of neurocognitive tests will be performed at baseline and 3 months post-SRS. Cognitive deterioration rate will be compared between the current trial and historical controls and linear regression used to analyze patient, tumor, and treatment related predictors of cognitive decline. Statistical modeling will be used to analyze changes in imaging biomarkers as a function of time and radiation dose, and these changes will be tested for association with domain-specific cognitive tests. Spatial sensitivity to RT dose across white matter tracts will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. One to three brain metastases targets, all smaller than 3 cm in diameter (intact or resected tumor bed)
3. Eastern cooperative Oncology Group (ECOG) performance status 0-2 (score of 0, no symptoms; 1, mild symptoms; 2, symptomatic, <50% in bed during the day)
4. Ability to answer questions and follow commands via neurocognitive testing
5. Estimated life expectancy greater than 6 months
6. Pathologic confirmation of extracerebral tumor site (eg, lung, breast, prostate) from either the primary site or a metastatic lesion
7. Willingness/Ability to undergo brain MRI scans
8. Able to give informed consent

Exclusion Criteria:

1. Pregnant or nursing women
2. Women of childbearing potential unwilling to use adequate contraception
3. Inability to complete a magnetic resonance imaging scan with contrast
4. Tumor directly invading the critical area to be spared (for example a patient with tumor invading a critical white matter tract; ineligible for cognitive-sparing)
5. Planned chemotherapy during SRS (on the day of SRS)
6. Previous whole brain radiation therapy
7. Leptomeningeal metastases (ineligible for SRS)
8. Metastases from primary germ cell tumor, small cell carcinoma, or primary CNS lymphoma (ineligible for SRS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Verbal Memory from baseline to 3 months after SRS | Change from Baseline (pre-treatment) to 3 months post treatment
  To evaluate the change from baseline to 3-month post-SRS verbal memory performance when performing relative sparing of eloquent white matter tracts and hippocampi from high doses during brain SRS in patients with 1 to 3 brain metastases. Verbal memory outcomes and measurements include: Hopkins Verbal Learning Test-Revised (HVLT-R)-Immediate, Delayed Recall. Scale of scores is 0-36 for Immediate, 0-12 for Delayed. For both tests, higher scores indicate better performance.
Change in Executive Functioning from baseline to 3 months after SRS | Change from Baseline (pre-treatment) to 3 months post treatment
  To evaluate the change from baseline to 3-month post-SRS executive functioning performance when performing relative sparing of eloquent white matter tracts and hippocampi from high doses during brain SRS in patients with 1 to 3 brain metastases. Executive functioning outcomes and measurements include: Controlled Oral Word Association Test (COWA): letter fluency, Trail Making Test Part B (TMT-B).
  Scale of scores is:
  Controlled Oral Word Association Test (COWA): letter fluency: 0- no upper limit. Higher score indicates better performance Trail Making Test Part B (TMT-B): 0-240. Higher score indicates poorer performance
Change in Attention/Processing Speed from baseline to 3 months after SRS | Change from Baseline (pre-treatment) to 3 months post treatment
  To evaluate the change from baseline to 3-month post-SRS Attention/Processing Speed performance when performing relative sparing of eloquent white matter tracts and hippocampi from high doses during brain SRS in patients with 1 to 3 brain metastases. Attention/Processing Speed outcomes and measurements include: Trail Making Test Part A (TMT-A)
  Scale of scores is:
  Trail Making Test Part A (TMT-A): 0-240. Higher score indicates poorer performance
Change in Language functioning from baseline to 3 months after SRS | Change from Baseline (pre-treatment) to 3 months post treatment
  To evaluate the change from baseline to 3-month post-SRS Language performance when performing relative sparing of eloquent white matter tracts and hippocampi from high doses during brain SRS in patients with 1 to 3 brain metastases. Language outcomes and measurements include: Boston Naming Test (BNT), Controlled Oral Word Association Test (COWA): category fluency
  Scale of scores is:
  Boston Naming Test (BNT): 0-60 Controlled Oral Word Association Test (COWA): category fluency: 0-no upper limit For both tests, higher score indicates better performance.

SECONDARY OUTCOMES:
Longitudinal changes in imaging biomarker fractional anisotropy (FA) from DTI imaging | baseline (pre-treatment), 3 months and 6 months post-treatment
  To measure longitudinal changes in FA (unitless index between 0 and 1) from DTI imaging
Longitudinal changes in imaging biomarker mean diffusivity (MD) from DTI imaging | baseline (pre-treatment), 3 months and 6 months post-treatment
  To measure longitudinal changes in MD (mm squared/second) from DTI imaging
Longitudinal changes in imaging biomarker volume from volumetric MR imaging | baseline (pre-treatment), 3 months and 6 months post-treatment
  To measure longitudinal changes in volume (cc) from volumetric MR imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jona Hattangadi-Gluth, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Moores Cancer Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arvold ND, Lee EQ, Mehta MP, Margolin K, Alexander BM, Lin NU, Anders CK, Soffietti R, Camidge DR, Vogelbaum MA, Dunn IF, Wen PY. Updates in the management of brain metastases. Neuro Oncol. 2016 Aug;18(8):1043-65. doi: 10.1093/neuonc/now127. PMID 27382120
- [Background] Nabors LB, Portnow J, Ammirati M, Baehring J, Brem H, Butowski N, Fenstermaker RA, Forsyth P, Hattangadi-Gluth J, Holdhoff M, Howard S, Junck L, Kaley T, Kumthekar P, Loeffler JS, Moots PL, Mrugala MM, Nagpal S, Pandey M, Parney I, Peters K, Puduvalli VK, Ragsdale J, Rockhill J, Rogers L, Rusthoven C, Shonka N, Shrieve DC, Sills AK, Swinnen LJ, Tsien C, Weiss S, Wen PY, Willmarth N, Bergman MA, Engh A. NCCN Guidelines Insights: Central Nervous System Cancers, Version 1.2017. J Natl Compr Canc Netw. 2017 Nov;15(11):1331-1345. doi: 10.6004/jnccn.2017.0166. PMID 29118226
- [Background] Scoccianti S, Detti B, Cipressi S, Iannalfi A, Franzese C, Biti G. Changes in neurocognitive functioning and quality of life in adult patients with brain tumors treated with radiotherapy. J Neurooncol. 2012 Jun;108(2):291-308. doi: 10.1007/s11060-012-0821-8. Epub 2012 Feb 18. PMID 22354791
- [Background] Greene-Schloesser D, Robbins ME. Radiation-induced cognitive impairment--from bench to bedside. Neuro Oncol. 2012 Sep;14 Suppl 4(Suppl 4):iv37-44. doi: 10.1093/neuonc/nos196. PMID 23095829
- [Background] Brown PD, Jaeckle K, Ballman KV, Farace E, Cerhan JH, Anderson SK, Carrero XW, Barker FG 2nd, Deming R, Burri SH, Menard C, Chung C, Stieber VW, Pollock BE, Galanis E, Buckner JC, Asher AL. Effect of Radiosurgery Alone vs Radiosurgery With Whole Brain Radiation Therapy on Cognitive Function in Patients With 1 to 3 Brain Metastases: A Randomized Clinical Trial. JAMA. 2016 Jul 26;316(4):401-409. doi: 10.1001/jama.2016.9839. PMID 27458945
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Lin NU, Wefel JS, Lee EQ, Schiff D, van den Bent MJ, Soffietti R, Suh JH, Vogelbaum MA, Mehta MP, Dancey J, Linskey ME, Camidge DR, Aoyama H, Brown PD, Chang SM, Kalkanis SN, Barani IJ, Baumert BG, Gaspar LE, Hodi FS, Macdonald DR, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Challenges relating to solid tumour brain metastases in clinical trials, part 2: neurocognitive, neurological, and quality-of-life outcomes. A report from the RANO group. Lancet Oncol. 2013 Sep;14(10):e407-16. doi: 10.1016/S1470-2045(13)70308-5. PMID 23993385
- [Background] Brown PD, Ballman KV, Cerhan JH, Anderson SK, Carrero XW, Whitton AC, Greenspoon J, Parney IF, Laack NNI, Ashman JB, Bahary JP, Hadjipanayis CG, Urbanic JJ, Barker FG 2nd, Farace E, Khuntia D, Giannini C, Buckner JC, Galanis E, Roberge D. Postoperative stereotactic radiosurgery compared with whole brain radiotherapy for resected metastatic brain disease (NCCTG N107C/CEC.3): a multicentre, randomised, controlled, phase 3 trial. Lancet Oncol. 2017 Aug;18(8):1049-1060. doi: 10.1016/S1470-2045(17)30441-2. Epub 2017 Jul 4. PMID 28687377
- [Background] Bagadia A, Purandare H, Misra BK, Gupta S. Application of magnetic resonance tractography in the perioperative planning of patients with eloquent region intra-axial brain lesions. J Clin Neurosci. 2011 May;18(5):633-9. doi: 10.1016/j.jocn.2010.08.026. Epub 2011 Mar 2. PMID 21371893
- [Background] Abhinav K, Yeh FC, Mansouri A, Zadeh G, Fernandez-Miranda JC. High-definition fiber tractography for the evaluation of perilesional white matter tracts in high-grade glioma surgery. Neuro Oncol. 2015 Sep;17(9):1199-209. doi: 10.1093/neuonc/nov113. Epub 2015 Jun 27. PMID 26117712
- [Background] Assaf Y, Pasternak O. Diffusion tensor imaging (DTI)-based white matter mapping in brain research: a review. J Mol Neurosci. 2008;34(1):51-61. doi: 10.1007/s12031-007-0029-0. PMID 18157658
- [Background] McDonald CR, Hagler DJ Jr, Girard HM, Pung C, Ahmadi ME, Holland D, Patel RH, Barba D, Tecoma ES, Iragui VJ, Halgren E, Dale AM. Changes in fiber tract integrity and visual fields after anterior temporal lobectomy. Neurology. 2010 Nov 2;75(18):1631-8. doi: 10.1212/WNL.0b013e3181fb44db. Epub 2010 Sep 29. PMID 20881271
- [Background] Cabezas M, Oliver A, Llado X, Freixenet J, Cuadra MB. A review of atlas-based segmentation for magnetic resonance brain images. Comput Methods Programs Biomed. 2011 Dec;104(3):e158-77. doi: 10.1016/j.cmpb.2011.07.015. Epub 2011 Aug 25. PMID 21871688
- [Background] Seibert TM, Karunamuni R, Bartsch H, Kaifi S, Krishnan AP, Dalia Y, Burkeen J, Murzin V, Moiseenko V, Kuperman J, White NS, Brewer JB, Farid N, McDonald CR, Hattangadi-Gluth JA. Radiation Dose-Dependent Hippocampal Atrophy Detected With Longitudinal Volumetric Magnetic Resonance Imaging. Int J Radiat Oncol Biol Phys. 2017 Feb 1;97(2):263-269. doi: 10.1016/j.ijrobp.2016.10.035. Epub 2016 Oct 31. PMID 28068234
- [Background] Connor M, Karunamuni R, McDonald C, White N, Pettersson N, Moiseenko V, Seibert T, Marshall D, Cervino L, Bartsch H, Kuperman J, Murzin V, Krishnan A, Farid N, Dale A, Hattangadi-Gluth J. Dose-dependent white matter damage after brain radiotherapy. Radiother Oncol. 2016 Nov;121(2):209-216. doi: 10.1016/j.radonc.2016.10.003. Epub 2016 Oct 21. PMID 27776747
- [Background] Connor M, Karunamuni R, McDonald C, Seibert T, White N, Moiseenko V, Bartsch H, Farid N, Kuperman J, Krishnan A, Dale A, Hattangadi-Gluth JA. Regional susceptibility to dose-dependent white matter damage after brain radiotherapy. Radiother Oncol. 2017 May;123(2):209-217. doi: 10.1016/j.radonc.2017.04.006. Epub 2017 May 2. PMID 28460824
- [Background] Seibert TM, Dalia Y, Karunamuni R, Piccioni D, McDonald CR, Farid N, Hattangadi-Gluth JA. Unilateral hippocampal wasting after combined-modality therapy for glioblastoma. Acta Oncol. 2018 May;57(5):688-691. doi: 10.1080/0284186X.2017.1398412. Epub 2017 Nov 10. No abstract available. PMID 29125006
- [Background] Gaspar L, Scott C, Rotman M, Asbell S, Phillips T, Wasserman T, McKenna WG, Byhardt R. Recursive partitioning analysis (RPA) of prognostic factors in three Radiation Therapy Oncology Group (RTOG) brain metastases trials. Int J Radiat Oncol Biol Phys. 1997 Mar 1;37(4):745-51. doi: 10.1016/s0360-3016(96)00619-0. PMID 9128946
- [Background] Johung KL, Yeh N, Desai NB, Williams TM, Lautenschlaeger T, Arvold ND, Ning MS, Attia A, Lovly CM, Goldberg S, Beal K, Yu JB, Kavanagh BD, Chiang VL, Camidge DR, Contessa JN. Extended Survival and Prognostic Factors for Patients With ALK-Rearranged Non-Small-Cell Lung Cancer and Brain Metastasis. J Clin Oncol. 2016 Jan 10;34(2):123-9. doi: 10.1200/JCO.2015.62.0138. Epub 2015 Oct 5. PMID 26438117
- [Background] Tsao MN, Rades D, Wirth A, Lo SS, Danielson BL, Gaspar LE, Sperduto PW, Vogelbaum MA, Radawski JD, Wang JZ, Gillin MT, Mohideen N, Hahn CA, Chang EL. Radiotherapeutic and surgical management for newly diagnosed brain metastasis(es): An American Society for Radiation Oncology evidence-based guideline. Pract Radiat Oncol. 2012 Jul-Sep;2(3):210-225. doi: 10.1016/j.prro.2011.12.004. Epub 2012 Jan 30. PMID 25925626
- [Background] Yamamoto M, Serizawa T, Shuto T, Akabane A, Higuchi Y, Kawagishi J, Yamanaka K, Sato Y, Jokura H, Yomo S, Nagano O, Kenai H, Moriki A, Suzuki S, Kida Y, Iwai Y, Hayashi M, Onishi H, Gondo M, Sato M, Akimitsu T, Kubo K, Kikuchi Y, Shibasaki T, Goto T, Takanashi M, Mori Y, Takakura K, Saeki N, Kunieda E, Aoyama H, Momoshima S, Tsuchiya K. Stereotactic radiosurgery for patients with multiple brain metastases (JLGK0901): a multi-institutional prospective observational study. Lancet Oncol. 2014 Apr;15(4):387-95. doi: 10.1016/S1470-2045(14)70061-0. Epub 2014 Mar 10. PMID 24621620
- [Background] Greene-Schloesser D, Robbins ME, Peiffer AM, Shaw EG, Wheeler KT, Chan MD. Radiation-induced brain injury: A review. Front Oncol. 2012 Jul 19;2:73. doi: 10.3389/fonc.2012.00073. eCollection 2012. PMID 22833841
- [Background] Gondi V, Pugh SL, Tome WA, Caine C, Corn B, Kanner A, Rowley H, Kundapur V, DeNittis A, Greenspoon JN, Konski AA, Bauman GS, Shah S, Shi W, Wendland M, Kachnic L, Mehta MP. Preservation of memory with conformal avoidance of the hippocampal neural stem-cell compartment during whole-brain radiotherapy for brain metastases (RTOG 0933): a phase II multi-institutional trial. J Clin Oncol. 2014 Dec 1;32(34):3810-6. doi: 10.1200/JCO.2014.57.2909. Epub 2014 Oct 27. PMID 25349290
- [Background] Gondi V, Tolakanahalli R, Mehta MP, Tewatia D, Rowley H, Kuo JS, Khuntia D, Tome WA. Hippocampal-sparing whole-brain radiotherapy: a "how-to" technique using helical tomotherapy and linear accelerator-based intensity-modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2010 Nov 15;78(4):1244-52. doi: 10.1016/j.ijrobp.2010.01.039. PMID 20598457
- [Background] Brown PD, Pugh S, Laack NN, Wefel JS, Khuntia D, Meyers C, Choucair A, Fox S, Suh JH, Roberge D, Kavadi V, Bentzen SM, Mehta MP, Watkins-Bruner D; Radiation Therapy Oncology Group (RTOG). Memantine for the prevention of cognitive dysfunction in patients receiving whole-brain radiotherapy: a randomized, double-blind, placebo-controlled trial. Neuro Oncol. 2013 Oct;15(10):1429-37. doi: 10.1093/neuonc/not114. Epub 2013 Aug 16. PMID 23956241
- [Background] Rapp SR, Case LD, Peiffer A, Naughton MM, Chan MD, Stieber VW, Moore DF Jr, Falchuk SC, Piephoff JV, Edenfield WJ, Giguere JK, Loghin ME, Shaw EG. Donepezil for Irradiated Brain Tumor Survivors: A Phase III Randomized Placebo-Controlled Clinical Trial. J Clin Oncol. 2015 May 20;33(15):1653-9. doi: 10.1200/JCO.2014.58.4508. Epub 2015 Apr 20. PMID 25897156
- [Background] Brown WR, Thore CR, Moody DM, Robbins ME, Wheeler KT. Vascular damage after fractionated whole-brain irradiation in rats. Radiat Res. 2005 Nov;164(5):662-8. doi: 10.1667/rr3453.1. PMID 16238444
- [Background] Wu PH, Coultrap S, Pinnix C, Davies KD, Tailor R, Ang KK, Browning MD, Grosshans DR. Radiation induces acute alterations in neuronal function. PLoS One. 2012;7(5):e37677. doi: 10.1371/journal.pone.0037677. Epub 2012 May 25. PMID 22662188
- [Background] Panagiotakos G, Alshamy G, Chan B, Abrams R, Greenberg E, Saxena A, Bradbury M, Edgar M, Gutin P, Tabar V. Long-term impact of radiation on the stem cell and oligodendrocyte precursors in the brain. PLoS One. 2007 Jul 11;2(7):e588. doi: 10.1371/journal.pone.0000588. PMID 17622341
- [Background] Monje ML, Mizumatsu S, Fike JR, Palmer TD. Irradiation induces neural precursor-cell dysfunction. Nat Med. 2002 Sep;8(9):955-62. doi: 10.1038/nm749. Epub 2002 Aug 5. PMID 12161748
- [Background] Koga T, Maruyama K, Kamada K, Ota T, Shin M, Itoh D, Kunii N, Ino K, Terahara A, Aoki S, Masutani Y, Saito N. Outcomes of diffusion tensor tractography-integrated stereotactic radiosurgery. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):799-802. doi: 10.1016/j.ijrobp.2010.11.046. Epub 2011 Jan 27. PMID 21277103
- [Background] Wang M, Ma H, Wang X, Guo Y, Xia X, Xia H, Guo Y, Huang X, He H, Jia X, Xie Y. Integration of BOLD-fMRI and DTI into radiation treatment planning for high-grade gliomas located near the primary motor cortexes and corticospinal tracts. Radiat Oncol. 2015 Mar 8;10:64. doi: 10.1186/s13014-015-0364-1. PMID 25884395
- [Background] Maruyama K, Koga T, Kamada K, Ota T, Itoh D, Ino K, Igaki H, Aoki S, Masutani Y, Shin M, Saito N. Arcuate fasciculus tractography integrated into Gamma Knife surgery. J Neurosurg. 2009 Sep;111(3):520-6. doi: 10.3171/2008.4.17521. PMID 19025357
- [Background] Zhang I, Antone J, Li J, Saha S, Riegel AC, Vijeh L, Lauritano J, Marrero M, Salas S, Schulder M, Zinkin H, Goenka A, Knisely J. Hippocampal-sparing and target volume coverage in treating 3 to 10 brain metastases: A comparison of Gamma Knife, single-isocenter VMAT, CyberKnife, and TomoTherapy stereotactic radiosurgery. Pract Radiat Oncol. 2017 May-Jun;7(3):183-189. doi: 10.1016/j.prro.2017.01.012. PMID 28477798
- [Background] Wang S, Wu EX, Qiu D, Leung LH, Lau HF, Khong PL. Longitudinal diffusion tensor magnetic resonance imaging study of radiation-induced white matter damage in a rat model. Cancer Res. 2009 Feb 1;69(3):1190-8. doi: 10.1158/0008-5472.CAN-08-2661. Epub 2009 Jan 20. PMID 19155304
- [Background] Peiffer AM, Shi L, Olson J, Brunso-Bechtold JK. Differential effects of radiation and age on diffusion tensor imaging in rats. Brain Res. 2010 Sep 10;1351:23-31. doi: 10.1016/j.brainres.2010.06.049. Epub 2010 Jul 1. PMID 20599817
- [Background] Zhu T, Chapman CH, Tsien C, Kim M, Spratt DE, Lawrence TS, Cao Y. Effect of the Maximum Dose on White Matter Fiber Bundles Using Longitudinal Diffusion Tensor Imaging. Int J Radiat Oncol Biol Phys. 2016 Nov 1;96(3):696-705. doi: 10.1016/j.ijrobp.2016.07.010. Epub 2016 Jul 21. PMID 27681767
- [Background] Chapman CH, Nagesh V, Sundgren PC, Buchtel H, Chenevert TL, Junck L, Lawrence TS, Tsien CI, Cao Y. Diffusion tensor imaging of normal-appearing white matter as biomarker for radiation-induced late delayed cognitive decline. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):2033-40. doi: 10.1016/j.ijrobp.2011.01.068. Epub 2011 May 11. PMID 21570218
- [Background] Chapman CH, Zhu T, Nazem-Zadeh M, Tao Y, Buchtel HA, Tsien CI, Lawrence TS, Cao Y. Diffusion tensor imaging predicts cognitive function change following partial brain radiotherapy for low-grade and benign tumors. Radiother Oncol. 2016 Aug;120(2):234-40. doi: 10.1016/j.radonc.2016.06.021. Epub 2016 Jul 11. PMID 27418525
- [Background] Heister D, Brewer JB, Magda S, Blennow K, McEvoy LK; Alzheimer's Disease Neuroimaging Initiative. Predicting MCI outcome with clinically available MRI and CSF biomarkers. Neurology. 2011 Oct 25;77(17):1619-28. doi: 10.1212/WNL.0b013e3182343314. Epub 2011 Oct 12. PMID 21998317
- See also: A Phase II Randomized Trial of Proton vs. Photon Therapy (IMRT) for Cognitive Preservation in Patients with IDH Mutant, Low to Intermediate Grade Gliomas. — https://www.nrgoncology.org/Clinical-Trials/Protocol-Table
- See also: A Randomized Phase III Trial of Memantine and Whole-Brain Radiotherapy With or Without Hippocampal Avoidance in Patients With Brain Metastases. — https://www.nrgoncology.org/Clinical-Trials/Protocol-Table

DOCUMENTS (1):
  • Study Protocol (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT04343157/Prot_000.pdf